CLINICAL TRIAL: NCT04195230
Title: Cognitive Training in a Multi-task Daily Life Task: a Feasibility Study in Healthy Older Adults
Brief Title: Cognitive Multi-Tasking Training in Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAS6529
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Age-related Cognitive Decline
Keywords: Web-based Cognitive Training; Executive Functions; Attention; Multi-tasking; Aging; Healthy Adults

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computerized Cognitive Training (Breakfast Game) (Experimental): Participants will undergo a pilot training protocol where they will have to perform two tasks concomitantly, in a multi-tasking fashion. The tasks are related to everyday activities as "cooking" and "setting tables".
  Interventions: Behavioral: Multi-tasking Training

INTERVENTIONS:
Behavioral: Multi-tasking Training — Participants will undergo training protocol where they will have, concomitantly, to cook different meals and set the table under different instructions, rules and difficulty level.

SUMMARY:
This study evaluated the feasibility of a remote web-based ecological cognitive training protocol to healthy older adults. The training protocol involves 5 training sessions.

DETAILED DESCRIPTION:
Previous research demonstrated the relevance in training cognitive abilities that typically decline with age, such as those associated with executive control (e.g., abstract thinking, selective and divided attention, planning, task-switching and inhibitory control). The aim of the present study is to investigate the feasibility of a web-based cognitive training focused on executive control to cognitively healthy older adults. The participants will undergo the web-training in a daily type situation of meal preparation (i.e., Breakfast Game). The training protocol combines the tasks of table setting and cooking in a multi-tasking fashion. In some sessions Emphasis Change approach will be apply to the training, in order to assess it feasibility and potential effects in optimizing the performance. In addition, participants will undergo a brief web-based cognitive evaluation before and after training. If feasible, the investigators protocol will allow training older adults in critical cognitive skills for daily life situations. The web-based training is an advancement since it can be delivered at-home, remotely supervised, and is easily scalable. Recently, remote interventions have been particularly relevant to older adults due to the COVID-19 pandemic, which may limit in-person research participation.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively healthy older adults

Exclusion Criteria:

* Low test scores (below 26 on the Montreal Cognitive Assessment - MoCA)
* Presence of certain medical conditions (i.e., major neurological or psychiatric disorder, or a medical condition that may impact cognitive functioning).
* Subjects which English is not the primary language, or with lack of capacity to consent will not be enrolled.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Change in Cooking Time Discrepancy Scores | Up to 3 weeks
  Change in cooking time (milliseconds) in each food type. In the computerized task, participants are asked to cook different food types. Scores reflect the average absolute values of the difference between the required and actual cooking time of each item. Lowers scores (closest to zero) represent a better outcome.
Change in Range of Stop Times Score | Up to 3 weeks
  Change in cooking time (milliseconds) between food items. In the computerized task, participants are asked to cook different food types. Scores reflect is the difference between the first and last food item stopped cooking. Lowers scores (closest to zero) represent a better outcome.
Change in the Number of Tables Set Score | Up to 3 weeks
  Change in the total number of tables set. In the computerized task, participants are asked to set tables for four guests, when finished, one point is given. Higher scores represent a better outcome.

SECONDARY OUTCOMES:
Post-training feasibility questionnaire | Within one week after the intervention
  Questionnaire assessing participant´s opinions about performing the web-based training based on Breakfast Game (e.g., difficulty, satisfaction). Higher scores reflect feasibility of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Yaakov Stern, Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by the principal investigator.

REFERENCES:
- [Derived] Sanz Simon S, Ben-Eliezer D, Pondikos M, Stern Y, Gopher D. Feasibility and acceptability of a new web-based cognitive training platform for cognitively healthy older adults: the breakfast task. Pilot Feasibility Stud. 2023 Aug 4;9(1):136. doi: 10.1186/s40814-023-01359-2. PMID 37542331